CLINICAL TRIAL: NCT02573844
Title: Efficacy of Proklama on Patients' Symptoms With Irritable Bowel Syndrome: Clinical Trial, Double- Blind, Crossover, Controlled Study vs. Placebo
Brief Title: Pain Relief In Irritable Bowel Syndrome
Acronym: PRITON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Geophyt S.r.l.s. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Geophyt
Record Dates: First submitted 2015-10-08; First posted 2015-10-12 (Estimated); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Irritable Bowel Syndrome
Keywords: irritable bowel syndrome; abdominal pain; rome III criteria; abdominal distension; consistency of stools; stool frequency; meteorism; flatulence; abdominal discomfort; proklama; probiotics; alga klamath; aphanizomenon flos-aquae; prebiotics; colitis ulcerosa
MeSH Terms: conditions — Irritable Bowel Syndrome; Abdominal Pain; Flatulence; Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: Proklama ( 1 sachet/ day) (Active Comparator): 15 patients belonging to group A will receive drug A (Proklama: 1 sachet/ day). The treatment will be administred starting from visit 3 for a 2 weeks- treatment's period.
  After a 2 weeks wash out's period, patients belonging to group A, starting from visit 5, will receive drug B ( Placebo: 1 sachet/day).
  Interventions: Drug: Proklama
- B: Placebo ( 1 sachet/ day) (Placebo Comparator): 15 patients belonging to group B will receive drug B (Placebo: 1 sachet/ day). The treatment will be administred starting from visit 3 for a 2 weeks- treatment's period.
  After a 2 weeks wash out's period, patients belonging to group B, starting from visit 5, will receive drug A ( Proklama: 1 sachet/day).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Proklama
  Arms: A: Proklama ( 1 sachet/ day)
Drug: Placebo
  Arms: B: Placebo ( 1 sachet/ day)

SUMMARY:
The purpose of this study is to determine whether Proklama is effective in significative reduction of pain, other symptoms IBS's related, and improves quality of life concerning IBS disease.

DETAILED DESCRIPTION:
This is a phase IV, double- blind, randomized, placebo controlled, monocentric study.

Males and women over 18 y.o. with Irritable bowel syndrome (IBS) diagnosed applying Rome III criteria will be enrolled consecutively.

The study consist of 4 periods:

* A screening's period of 2 weeks starting from visit 1, useful to screen potentially eligible patients performing diagnostic investigations necessary to confirm diagnosis.
* A run- in's period, starting from visit 2 and lasting 2 weeks will represent a baseline without specific treatments in order to characterize the severity of symptomatology and evaluate patients' compliance relative to daily diaries
* A 2 weeks- treatment's period ( active/ placebo) starting from visit 3. The 1st day of the period of treatment, eligible patients will be randomized following a 1:1 ratio to receive Proklama ( 1 sachet/ day) or placebo. Treatments will be administered daily during the whole 2 weeks- treatment's period.
* A wash out's period lasting 2 weeks starting from visit 4, to be performed the day after the end of the 2 weeks- treatment's period.
* A 2 weeks- treatment's period ( placebo/ active) starting from visit 5, to be performed the last day of wash out's period. During this visit patients will receive the second treatment, following a crossover design.

ELIGIBILITY:
Inclusion Criteria:

1. patients over 18 y.o.
2. clinical diagnosis of IBS following Rome III symptom- based criteria:

   1. abdominal pain or discomfort recurring for at least 3 days a month in the previous 3 months, associated with 2 of the following characteristics at least: improved with evacuation; onset associated with variation of stool frequency; onset associated with changes in stool consistency
   2. onset of symptomatology at least 6 months preceding diagnosis
   3. additional criterion: mean severity of abdominal pain higher than 3 in the 11-points NRS
3. For patients over 50 y.o. or with positive familiarity for colorectal cancer: normal colonoscopy performed within 5 years from the beginning of the screening's period and after symptomatology's onset
4. For patients over 65 y.o. : absence of ischemic / microscopic colitis, or other organic gastrointestinal disorders, as highlighted through colonoscopy with biopsy performed within 6 months from the beginning of the screening's period
5. For fertile and sexually active women: use of effective contraception with failure rate of less than 1% for one year during the trial period and 30 days after its end.

   Oral contraceptive are admitted as long as formulation didn't undergo changes during the 6 months preceeding the trial.
6. Physical examination is negative during the period of screening
7. Absence of significant alterations in 12- lead ECG during the period of screening.
8. Normal haematochemical parameters during the period of screening
9. Compliant patients towards procedures provided for the study, especially the use of daily diary
10. Patients with mental integrity, able to express an informed before any procedure related to protocol, compliant toward clinical examinations provided for the protocol.
11. Patients willing to avoid loperamide and laxatives use during the 3 days preceding run in and during the whole run in's period ( to be verified before randomization)
12. Patients that during both the 2 run in's weeks reported an average daily intensity of abdominal pain for every week >3 on 0-10 (NRS)

Exclusion Criteria:

1. Male gender
2. Patient has a diagnosis of IBS with a subtype of constipation, mixed IBS, or unsubtyped IBS according to the Rome III criteria
3. Patient has had surgery that meets any of the following criteria:

   a) colonic or major abdominal surgery, i.e. bariatric surgery and stomach, small/ large bowel or large vessel abdominal surgery ( except appendicectomy, hysterectomy, cholecystectomy, caesarean section, or laparoscopic surgery).
4. Patient has any elective major surgery planned or expected at any time during the study.
5. Patient has a history of inflammation bowel diseases, complicated diverticulosis ( i.e. diverticulitis), ischaemic colitis, microscopic colitis.
6. Patient has a history of organic abnormalities of the GI tract, intestinal obstruction, stricture, toxic megacolon, GI perforation, fecal impaction, gastric banding, adhesions or impaired intestinal circulation ( e.g., aortoiliac disease).
7. Patient has a history of pancreatitis of any etiology, cholecystitis or of symptomatic gallbladder stone disease in the previous 6 months.
8. Patient has an active biliary duct disease of a history of Sphincter of Oddi dysfunction.
9. Patient has a history of gluten enteropathy.
10. Patient has a history of lactose intolerance as assessed by response to diet.
11. Patient has a current or previous diagnosis of neoplasia ( except non-GI) neoplasia in complete remission < or = 5 years, squamous and basal cell carcinomas and cervical carcinoma in situ).
12. Patient has a history of ectopic endometriosis.
13. Patient has a history of positive tests for ova or parasites, or clostridium difficile toxin or occult blood in the stool in the previous 6 months.
14. Patient has a history of human immunodeficiency virus infection.
15. Patient has a history of a cardiovascular event, including stroke, myocardial infarction, congestive heart failure ( NYHA class > 2), or transient ischemic attack in the previous 6 months.
16. Patient has uncontrolled hypertension, defined as systolic blood pressure <180 mmHg or a diastolic blood pressure < 100 mmHg.
17. Patient has insulin- dependent diabetes mellitus.
18. Patient has a major pshychiatric or neurological disorders.
19. Patient has an unstable medical condition which may compromise the efficacy and safety assessments as required in the study and/or require change in concomitant medication.
20. Patient has a history of abnormal thyroid function. Patient is candidate for the study if thyroid hormone replacement therapy is stable from at least 2 months.
21. Patient has evidence of clinically hepatic disease as defined by alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 times rthe upper limit of normal or total bilirubin >3 mg/dl (>51.3 mmoL/L), with the exception of Gilbert's syndrome or albumin < 2.8 g/dL during the Screening period.
22. Patient has a sever renal insufficiency ( Glomerular Filtration Rate [GFR] <30 mL/min/ 1.73 m^2 calculated by the Cockcroft. Gault formula adjusted for the body surface area [BSA]) during the Screening period
23. Patient has evidence of anemia as confirmed by hemoglobin < 9 g/dL during the Screening period.
24. Relevant changes in dietary habits, lifestyle or exercise regimen should be maintained for the duration of the study.
25. Use of prohibited concurrent medication within the previous month, namely:

    * Antibiotics ( 4 months in the case of rifaximin);
    * 5- HT3 antagonists alosetron.
26. Use of prohibited concurrent medication in the previous 7 days namely:

    * Antimuscarinic drugs;
    * Drug enhancing GI motility such as prokinetic agents and other stimulants of GI contractility drugs, laxatives, or anti- diarrhoeal agents ( except for loperamide, please refer to inclusion criterion No.12);
    * Analgesic drugs ( opioids or non- steroidal anti- inflammatory drugs). NOTE: short term use of paracetamol is allowed for max 2 consecutive days;
    * Fibre products and herbal preparations;
    * Antidepressants. NOTE: the use of a single antidepressant is only allowed when the drug type and its dose regimen have not been changed in the previous 6 months;
    * Benzodiazepines. NOTE: the use of a single benzodiazepine is only allowed when it is administered as sleep- inducer and the drug type and its dose regimen have not been changed in the previous 6 months.
27. Pregnancy or breastfeeding.
28. Hypersensitivity to the drug excipients.
29. Patient is not able to understand or collaborate throughout the study.
30. Patient is unable to swallow solid, oral dosage forms whole with the aid of liquid ( patients may not chew, divide, dissolve, or crush the study drug).
31. Partecipation in other clinical studies in the previous 4 weeks or the patient is currently enrolled in a clinical study with another investigational drug.
32. Patient has any condition that, in the opinion of the Investigator, would compromise the well- being of the patient or the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01; Primary Completion 2017-10 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Recorded pain in a diary using a 11-points Numeric Rating Scale (NRS) | 24 h
  Self reported evaluation of the most severe pain occurred in the previous 24 hours.
  Pain severity is scored 0-10 ( 0= absent; 10= pain as bad as can be).

SECONDARY OUTCOMES:
Recorded abdominal distension in a diary using a 11-points Numeric Rating Scale (NRS) | 24 h
  Self reported evaluation of abdominal distension occurred in the previous 24 hours.
  Abdominal distension is scored 0-10 ( 0= absent; 10= abdominal distension as bad as can be).
Recorded abdominal discomfort in a diary using a 11-points Numeric Rating Scale (NRS) | 24 h
  Self reported evaluation of abdominal discomfort occurred in the previous 24 hours.
  Abdominal discomfort is scored 0-10 ( 0= absent; 10= abdominal discomfort as bad as can be).
Recorded abdominal meteorism in a diary using a 11-points Numeric Rating Scale (NRS) | 24 h
  Self reported evaluation of abdominal meteorism occurred in the previous 24 hours.
  Abdominal meteorism is scored 0-10 ( 0= absent; 10= abdominal meteorism as bad as can be).
Recorded flatulence in a diary using a 11-points Numeric Rating Scale (NRS) | 24 h
  Self reported evaluation of flatulence occurred in the previous 24 hours. Flatulence is scored 0-10 ( 0= absent; 10= flatulence as bad as can be).
Recorded borborygmi in a diary using a 11-points Numeric Rating Scale (NRS) | 24 h
  Self reported evaluation of borgorygms occurred in the previous 24 hours. Borborygmi is scored 0-10 ( 0= absent; 10= borborygmi as bad as can be).
Recorded nausea in a diary using a 11-points Numeric Rating Scale (NRS) | 24 h
  Self reported evaluation of nausea occurred in the previous 24 hours. Nausea is scored 0-10 ( 0= absent; 10= nausea as bad as can be).
Recorded belching in a diary using a 11-points Numeric Rating Scale (NRS) | 24 h
  Self reported evaluation of belching occurred in the previous 24 hours. Belching is scored 0-10 ( 0= absent; 10= belching as bad as can be).
Recorded asthenia in a diary using a 11-points Numeric Rating Scale (NRS) | 24 h
  Self reported evaluation of asthenia occurred in the previous 24 hours. Asthenia is scored 0-10 ( 0= absent; 10= asthenia as bad as can be).
Recorded headache in a diary using a 11-points Numeric Rating Scale (NRS) | 24 h
  Self reported evaluation of headache occurred in the previous 24 hours. Headache is scored 0-10 ( 0= absent; 10= headache as bad as can be).
Recorded "empty- head" feeling in a diary using a 11-points Numeric Rating Scale (NRS) | 24 h
  Self reported evaluation of "empty- head" feeling occurred in the previous 24 hours.
  "Empty- head" feeling is scored 0-10 ( 0= absent; 10= "empty- head" feeling as bad as can be).
Recorded attention deficity in a diary using a 11-points Numeric Rating Scale (NRS) | 24 h
  Self reported evaluation of attention deficity occurred in the previous 24 hours.
  Attention deficity is scored 0-10 ( 0= absent; 10= attention deficity as bad as can be).
Recorded vomiting feeling in a diary using a 11-points Numeric Rating Scale (NRS) | 24 h
  Self reported evaluation of vomiting occurred in the previous 24 hours. Vomiting feeling is scored 0-10 ( 0= absent; 10= vomiting as bad as can be).
Recorded heartburn in a diary using a 11-points Numeric Rating Scale (NRS) | 24 h
  Self reported evaluation of heartburn occurred in the previous 24 hours. Heartburn is scored 0-10 ( 0= absent; 10= heartburn as bad as can be).
Number of evacuations recorded in a diary | 24 h
  Self reported record of number of evacuations in the previous 24 h.
Recorded stool consistency in a diary using a 7- point Bristol Stool Form Scale | 24 h
  Self reported evaluation of stool consistency occurred in the previous 24 hours.
  Stool consistency is scored 1- 7 ( 1= constipation; 7=diarrhoea)

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico San Matteo Pavia Fondazione IRCCS, Pavia, Italy